CLINICAL TRIAL: NCT05341414
Title: Resilience Trajectories Following a Preoperative Lifestyle /Behavioral Modification Program and Bariatric Surgery
Brief Title: Trajectories of Resilience and Bariatric Surgery Outcomes
Acronym: ECLAIRCIE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Olivier ZIEGLER, Clinical Professor, Central Hospital, Nancy, France
Other Study IDs: 2020PI203
Record Dates: First submitted 2022-03-21; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Severe Obesity; Psychological Distress; Bariatric Surgery Candidate
Keywords: Severe obesity; Resilience; Trauma; Psychological disorders; Eating disorders; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Wounds and Injuries; Mental Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A high prevalence of psychological trauma on one hand and of psychiatric disorders, such as depression, anxiety, suicide attempts, addictions, and eating disorders on the other hand, has been reported in patients with severe obesity seeking bariatric surgery. Some studies reported an increased prevalence of these psychiatric disorders after bariatric surgery, potentially related to weight regain. In this context, psychological resilience is a concept that brings together internal and external factors of adaptation, and whose clinical use facilitates interdisciplinary collaborative work. This research focuses on the association between resilience and success or failure of bariatric surgery in patients followed in the Specialized Obesity Center (CSO) of the Nancy University Hospital. The hypothesis is that psychological resilience before surgery promotes successful surgical treatment. This retrospective study is based on existing data from patients with severe obesity who have undergone bariatric surgery at the Nancy CSO. The main objective is to study 1) the resilience of patients with severe obesity, candidates for bariatric surgery, at the first assessment (T0), at the end of lifestyle/behavioral modifications program (T1) and at 2 years after bariatric surgery (T2), 2) the relationship between internal and external factors explaining resilience and final weight outcomes.

The investigators are expected that non-resilient patients have more psychological vulnerabilities (psychopathology, negative life events, etc.), and have lower weight loss than resilient patients.

DETAILED DESCRIPTION:
The investigators will report the change of resilience during lifestyle/behavioral modifications program and 2 years after bariatric surgical treatment, and the investigators will describe the factors associated with this change:

* History of trauma
* Psychopathology (eating disorders, depression, anxiety, addiction)
* Personality factors
* Characteristic of psychotherapy

ELIGIBILITY:
Inclusion Criteria:

* Severe obesity (BMI ≥35 kg/m2)
* Candidate for Bariatric surgery at Nancy CSO (2016-2020) after a lifestyle/behavioral modifications program
* Full psychological assessment data

Exclusion Criteria:

* Patient's opposition to the use of data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking for bariatric surgery at the Nancy CSO
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Resilience (Questionnaire) : Resilience Scale for Adult (RSA) | baseline (T0)
  Min: 33 ; Max: 231; Higher scores mean a better outcome Score of resilience (Resilience Scale for adults) and level of resilience (non-resilient, intermediate, resilient) / number of patients in each category
Resilience (semi-structured interview) : level of resilience | baseline (T0)
  Categories : Non-resilient, intermediate, resilient Number and % of patients in each category
Resilience (Questionnaire) : Resilience Scale for Adult (RSA) | 10 months (T1)
  Min: 33 ; Max: 231; Higher scores mean a better outcome
Resilience (semi-structured interview) : level of resilience | 10 months (T1)
  Categories : Non-resilient, intermediate, resilient Number and % of patients in each category
Resilience (Questionnaire) : Resilience Scale for Adult (RSA) | 2 years after surgery (T2)
  Min: 33 ; Max: 231; Higher scores mean a better outcome.
Resilience (semi-structured interview) : level of resilience | 2 years after surgery (T2)
  Categories : Non-resilient, intermediate, resilient Number and % of patients in each category

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale (HAD) | baseline (T0)
  Min: 0 ; Max: 42; Higher scores mean a worse outcome.
Dutch Eating Behaviour Questionnaire (DEBQ) | baseline (T0)
  Min: 33 ; Max: 165 ; Higher scores mean a worse outcome
Binge eating scale (BES) | baseline (T0)
  Min: 0 ; Max: 48 ; Higher scores mean a worse outcome.
Mini International Neuropsychiatric Interview (semi-structured interview) | baseline (T0)
  Number and % of patients in each category (major depressive episode, dysthymia, suicidal risk, bipolar disorder, panic disorder, agoraphobia, social phobia, obsessive compulsive disorder, post-traumatic stress disorders, alcohol (addiction/abuse), drugs (addiction/abuse), psychotic disorders, generalized anxiety, anti- social personality disorders, eating disorders).
Psychological trauma (semi-structured interview) | Baseline (T0)
  Number and % of patients in each category (Sexual, physical, emotional abuse, emotional and physical neglect) Number and % of patients in each category for the first trauma (childhood, adolescence, adulthood)
Childhood Trauma Questionnaire (CTQ) | baseline (T0)
  Min: 25 ; Max: 125 ; Higher scores mean a worse outcome
Toronto Alexithymia Scale (TAS) | baseline (T0)
  Min: 20 ; Max: 100 ; Higher scores mean a worse outcome
Medical Outcomes Study Short Form (SF-36) | baseline (T0)
  Min: 0 ; Max: 100 ; Higher scores mean a better outcome.
Definition of patient's psychological profile : clinical interviews | baseline (T0)
  Profile is determined by clinical interviews
Definition of patient's psychological profile : Rorschach test | baseline (T0)
  Profile is determined by Rorschach test
Characteristics of psychotherapy : Duration | baseline (T0)
  Duration of psychotherapy (month)
Characteristics of psychotherapy : Frequency | baseline (T0)
  Frequency of psychotherapy (number of sessions per month)
Characteristics of psychotherapy: Type of professional | baseline (T0)
  Type of professional (Psychiatrist, Psychologist, Nurse, Other)
Characteristics of psychotherapy : Investment | baseline (T0)
  Investment in psychotherapy (0:bad ; 5: excellent) Min: 0 ; Max: 5 ; Higher scores mean a better outcome.
Sex | baseline (T0)
  men/women
Age | baseline (T0)
  years
Professional situation | baseline (T0)
  Active / Unemployed / Homemaker / Retired / Unable to work
Family situation | baseline (T0)
  Currently married/cohabiting / Formerly married / Never married
Weight data | baseline (T0)
  Weight: kg BMI: kg/m²
Hospital Anxiety and Depression scale (HAD) | 10 months (T1)
  Min: 0 ; Max: 42; Higher scores mean a worse outcome
Dutch Eating Behaviour Questionnaire (DEBQ) | 10 months (T1)
  Min: 33 ; Max: 165 ; Higher scores mean a worse outcome
Binge eating scale (BES) | 10 months (T1)
  Min: 0 ; Max: 48 ; Higher scores mean a worse outcome
Mini International Neuropsychiatric Interview | 10 months (T1)
  • Number and % of patients in each category (major depressive episode, dysthymia, suicidal risk, bipolar disorder, panic disorder, agoraphobia, social phobia, obsessive compulsive disorder, post-traumatic stress disorders, alcohol (addiction/abuse), drugs (addiction/abuse), psychotic disorders, generalized anxiety, anti- social personality disorders, eating disorders).
Toronto Alexithymia Scale (TAS) | 10 months (T1)
  Min: 20 ; Max: 100 ; Higher scores mean a worse outcome.
Medical Outcomes Study Short Form (SF-36) | 10 months (T1)
  Min: 0 ; Max: 100 ; Higher scores mean a better outcome.
Definition of patient's psychological profile :clinical interviews | 10 months (T1)
  Profile is determined by clinical interviews
Definition of patient's psychological profile : Rorschach test | 10 months (T1)
  Profile is determined by Rorschach test
Characteristics of psychotherapy: Duration | 10 months (T1)
  Duration of psychotherapy (month)
Characteristics of psychotherapy: Frequency | 10 months (T1)
  Frequency of psychotherapy (number of sessions per month)
Characteristics of psychotherapy: Type of professional | 10 months (T1)
  Type of professional (Psychiatrist, Psychologist, Nurse, Other)
Characteristics of psychotherapy: Investment | 10 months (T1)
  Investment in psychotherapy (0:bad ; 5: excellent) Min: 0 ; Max: 5 ; Higher scores mean a better outcome.
Professional situation | 10 months (T1)
  Active / Unemployed / Homemaker / Retired / Unable to work
Family situation | 10 months (T1)
  Currently married/cohabiting / Formerly married / Never married
Weight data | 10 months (T1)
  Weight: kg BMI: kg/m²
Hospital Anxiety and Depression scale (HAD) | 2 years after surgery (T2)
  Min: 0 ; Max: 42; Higher scores mean a worse outcome.
Dutch Eating Behaviour Questionnaire (DEBQ) | 2 years after surgery (T2)
  Min: 33 ; Max: 165 ; Higher scores mean a worse outcome.
Binge eating scale (BES) | 2 years after surgery (T2)
  Min: 0 ; Max: 48 ; Higher scores mean a worse outcome.
Mini International Neuropsychiatric Interview | 2 years after surgery (T2)
  • Number and % of patients in each category (major depressive episode, dysthymia, suicidal risk, bipolar disorder, panic disorder, agoraphobia, social phobia, obsessive compulsive disorder, post-traumatic stress disorders, alcohol (addiction/abuse), drugs (addiction/abuse), psychotic disorders, generalized anxiety, anti- social personality disorders, eating disorders).
Toronto Alexithymia Scale (TAS) | 2 years after surgery (T2)
  Min: 20 ; Max: 100 ; Higher scores mean a worse outcome.
Medical Outcomes Study Short Form (SF-36) | 2 years after surgery (T2)
  Min: 0 ; Max: 100 ; Higher scores mean a better outcome.
Definition of patient's psychological profile : clinical interviews | 2 years after surgery (T2)
  Profile is determined by clinical interviews
Definition of patient's psychological profile : Rorschach test | 2 years after surgery (T2)
  Profile is determined by Rorschach test
Characteristics of psychotherapy: Duration | 2 years after surgery (T2)
  Duration of psychotherapy (month)
Characteristics of psychotherapy: Frequency | 2 years after surgery (T2)
  Frequency of psychotherapy (number of sessions per month)
Characteristics of psychotherapy: Type of professional | 2 years after surgery (T2)
  Type of professional (Psychiatrist, Psychologist, Nurse, Other)
Characteristics of psychotherapy: Investment | 2 years after surgery (T2)
  Investment in psychotherapy (0:bad ; 5: excellent) Min: 0 ; Max: 5 ; Higher scores mean a better outcome.
Professional situation | 2 years after surgery (T2)
  Active / Unemployed / Homemaker / Retired / Unable to work
Family situation | 2 years after surgery (T2)
  Currently married/cohabiting / Formerly married / Never married
Weight data | 2 years after surgery (T2)
  Weight: kg BMI: kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Ziegler, PU-PH, Principal Investigator — CHRU -Nancy, Université de Lorraine
Locations (1):
- Centre hospitalo-universitaire régional de Nancy, Vandœuvre-lès-Nancy, France